CLINICAL TRIAL: NCT02193867
Title: A Phase 2, Open Label, Multicenter Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Sebelipase Alfa in Infants With Rapidly Progressive Lysosomal Acid Lipase Deficiency
Brief Title: Clinical Study In Infants With Rapidly Progressive Lysosomal Acid Lipase Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-CL08
Record Dates: First submitted 2014-07-07; First posted 2014-07-18 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: LIPA; Wolman Disease; Wolman Phenotype; Acid Lipase Deficiency; Acid Cholesteryl Hydrolase; Acid Lipase Disease Deficiency, type 2; Cholesteryl Ester Storage Disease (CESD); Cholesteryl Ester Hydrolase Deficiency; Early Onset Lysosomal Acid Lipase Deficiency (Wolman Disease); LAL Deficiency; Late Onset Lysosomal Acid Lipase Deficiency (CESD); Wolman Disease (early onset LAL Deficiency); Related Disorders:; Non-alcoholic Fatty Liver Disease (NAFLD); Non-alcoholic Steatohepatitis (NASH); Alcoholic Liver Disease; Cryptogenic Cirrhosis; Niemann-Pick Disease (NPD) Type C; Chanarin Dorfman Syndrome
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease; Non-alcoholic Fatty Liver Disease; Liver Diseases, Alcoholic; Cirrhosis, Cryptogenic; Niemann-Pick Diseases; Chanarin-Dorfman Syndrome | interventions — Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Sebelipase Alfa (Experimental): All participants initiated once weekly (qw) intravenous (IV) infusions with sebelipase alfa at a dose of 1 milligram/kilogram (mg/kg) qw. A participant who met protocol defined dose escalation criteria at a dose of 1 mg/kg qw could be considered for a dose escalation to 3 mg/kg qw. If a participant continued to meet dose escalation criteria after at least 4 infusions at a dose of 3 mg/kg qw, the participant could be considered for a further dose escalation to 5 mg/kg qw. Under country-specific provisions (United Kingdom only), participants could be considered for a further dose escalation to 7.5 mg/kg qw if a thorough case review indicated that a participant continued to have evidence of disease progression at a dose of 5 mg/kg qw. All dose escalations were contingent upon acceptable safety and tolerability of preceding infusions and were undertaken by mutual agreement of the Investigator and Sponsor and after approval by an independent safety committee.
  Interventions: Drug: Sebelipase Alfa

INTERVENTIONS:
Drug: Sebelipase Alfa — Sebelipase alfa is a recombinant human lysosomal acid lipase. The investigational medicinal product is an enzyme replacement therapy intended for treatment of participants with LAL-D. Dosing occurred once weekly for up to 3 years.
  Other Names: SBC-102

SUMMARY:
This was an open-label, repeat-dose, study of sebelipase alfa in infants with rapidly progressive lysosomal acid lipase deficiency (LAL-D). Eligible participants received once-weekly infusions of sebelipase alfa for up to 3 years.

DETAILED DESCRIPTION:
Lysosomal acid lipase deficiency is a rare autosomal recessive lipid storage disorder that is caused by a marked decrease or complete absence of the LAL enzyme, leading to the accumulation of lipids, predominately cholesteryl esters and triglycerides, in various tissues and cell types. In the liver, accumulation of lipids in hepatocytes and macrophages leads to hepatomegaly, fibrosis, cirrhosis, liver dysfunction, and hepatic failure. In the small intestine, lipid-laden macrophage accumulation in the lamina propria leads to profound malabsorption.

Lysosomal acid lipase deficiency presenting in infancy is an extremely rare form of the disease characterized by profound malabsorption, growth failure, and hepatic failure that is usually fatal within the first 6 months of life.

ELIGIBILITY:
Inclusion Criteria:

1. Participant's parent or legal guardian (if applicable) consent to participation in the study
2. Confirmation of documented decreased LAL activity relative to the normal range of the lab performing the assay or confirmation of LAL-D diagnosis as determined by a Sponsor-approved central laboratory
3. Substantial clinical concerns, in the opinion of Investigator and Sponsor, of rapid disease progression requiring urgent medical intervention including, but not restricted to the following:

   * Marked abdominal distension and hepatomegaly
   * Failure to thrive
   * Disturbance of coagulation
   * Severe anemia
   * Sibling with rapidly progressive course of LAL-D

Exclusion Criteria:

1. Clinically important concurrent disease
2. Participant was > 8 months of age at the time of first dosing
3. Participant received an investigational medicinal product other than sebelipase alfa within 14 days prior to the first dose of sebelipase alfa in this study
4. Myeloablative preparation, or other systemic pre-transplant conditioning, for hematopoietic stem cell or liver transplantation
5. Previous hematopoietic stem cell or liver transplant
6. Known hypersensitivity to eggs

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Phoenix, Arizona, United States
- Kuopio, Finland
- Naples, Italy
- United Kingdom (2):
  - Birmingham
  - Manchester

REFERENCES:
- [Background] Balwani M, Breen C, Enns GM, Deegan PB, Honzik T, Jones S, Kane JP, Malinova V, Sharma R, Stock EO, Valayannopoulos V, Wraith JE, Burg J, Eckert S, Schneider E, Quinn AG. Clinical effect and safety profile of recombinant human lysosomal acid lipase in patients with cholesteryl ester storage disease. Hepatology. 2013 Sep;58(3):950-7. doi: 10.1002/hep.26289. Epub 2013 Mar 28. PMID 23348766
- [Background] Jones SA, Valayannopoulos V, Schneider E, Eckert S, Banikazemi M, Bialer M, Cederbaum S, Chan A, Dhawan A, Di Rocco M, Domm J, Enns GM, Finegold D, Gargus JJ, Guardamagna O, Hendriksz C, Mahmoud IG, Raiman J, Selim LA, Whitley CB, Zaki O, Quinn AG. Rapid progression and mortality of lysosomal acid lipase deficiency presenting in infants. Genet Med. 2016 May;18(5):452-8. doi: 10.1038/gim.2015.108. Epub 2015 Aug 27. PMID 26312827
- [Background] Jones SA, Rojas-Caro S, Quinn AG, Friedman M, Marulkar S, Ezgu F, Zaki O, Gargus JJ, Hughes J, Plantaz D, Vara R, Eckert S, Arnoux JB, Brassier A, Le Quan Sang KH, Valayannopoulos V. Survival in infants treated with sebelipase Alfa for lysosomal acid lipase deficiency: an open-label, multicenter, dose-escalation study. Orphanet J Rare Dis. 2017 Feb 8;12(1):25. doi: 10.1186/s13023-017-0587-3. PMID 28179030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 sites were initiated, and participants were treated at 5 sites in 4 countries (United Kingdom [UK], United States [US], Finland, Italy). One study site in the US was initiated but did not screen or treat any participants.
Pre-assignment Details: The study consisted of a screening period of up to 3 weeks. Participants who met all eligibility criteria were enrolled, treated, and analyzed.
Groups:
- Open-Label Sebelipase Alfa: All participants initiated once weekly (qw) intravenous (IV) infusions with sebelipase alfa at a dose of 1 milligram/kilogram (mg/kg) qw. A participant who met protocol defined dose escalation criteria at a dose of 1 mg/kg qw could be considered for a dose escalation to 3 mg/kg qw. If a participant continued to meet dose escalation criteria after at least 4 infusions at a dose of 3 mg/kg qw, the participant could be considered for a further dose escalation to 5 mg/kg qw. Under country-specific provisions (UK only), participants could be considered for a further dose escalation to 7.5 mg/kg qw if a thorough case review indicated that a participant continued to have evidence of disease progression at a dose of 5 mg/kg qw. All dose escalations were contingent upon acceptable safety and tolerability of preceding infusions and were undertaken by mutual agreement of the Investigator and Sponsor and after approval by an independent safety committee.
Period: Overall Study
Arm/Group | Open-Label Sebelipase Alfa
Started | 10
Received At Least 1 Dose Of Study Drug (Full Analysis Set (FAS)) | 10
Completed 18 Months Of Treatment (Treatment was to be at least 18 months; participants could continue treatment for up to 3 years) | 8
Completed (All participants continued to receive commercial therapy after study completion/Sponsor termination) | 6
Not Completed | 4
Not completed — Death | 2
Not completed — Sponsor Study Termination | 2

BASELINE CHARACTERISTICS:
Population: FAS: All participants who received any amount of sebelipase alfa (1.0, 3.0, 5.0, or 7.5 mg/kg qw) during the study.
Groups:
- Open-Label Sebelipase Alfa: All participants initiated qw IV infusions with sebelipase alfa at a dose of 1 mg/kg qw. A participant who met protocol defined dose escalation criteria at a dose of 1 mg/kg qw could be considered for a dose escalation to 3 mg/kg qw. If a participant continued to meet dose escalation criteria after at least 4 infusions at a dose of 3 mg/kg qw, the participant could be considered for a further dose escalation to 5 mg/kg qw. Under country-specific provisions (UK only), participants could be considered for a further dose escalation to 7.5 mg/kg qw if a thorough case review indicated that a participant continued to have evidence of disease progression at a dose of 5 mg/kg qw. All dose escalations were contingent upon acceptable safety and tolerability of preceding infusions and were undertaken by mutual agreement of the Investigator and Sponsor and after approval by an independent safety committee.
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.13 (2.859)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 1
  Race/Ethnicity: Asian | 6
  Race/Ethnicity: White | 1
  Race/Ethnicity: Egyptian | 1
  Race/Ethnicity: Turkish Kurdish | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Severe Treatment-emergent Adverse Events (TEAEs)
Description: The number of participants experiencing severe TEAEs is presented for participants who received sebelipase alfa in this open-label study. Adverse events were obtained through spontaneous reporting or elicited by specific questioning or examination of the participant's parent or legal guardian. An adverse event was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant, whether or not causally related to administration of study drug. Adverse event severity was graded by the Investigator as mild, moderate, or severe based on definitions developed from Clinical Data Interchange Standards Consortium Study Data Tabulation Model standard terminology v3.1.1. Adverse events reporting was from the date of informed consent until completion of the follow-up visit at approximately 30 days after the last dose of study drug. A summary of all serious and other nonserious AEs regardless of causality is located in the Reported AE module.
Time Frame: Screening through Month 37
Population: FAS: All participants who received any amount of sebelipase alfa (1.0, 3.0, 5.0, or 7.5 mg/kg qw) during the study and where applicable, met end point criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Percentage Of Participants Surviving To 12, 18, 24, And 36 Months Of Age
Description: The percentage of participants in the FAS who survived to 12, 18, 24, and 36 months of age. The exact confidence interval was calculated using the Clopper-Pearson method. Participants with unknown survival status at the age specified in the analysis were excluded. At 36 months, there were 2 participants who were alive and still on study who had not yet reached the age specified in the analysis. As such, these participants were excluded from the calculation of percent surviving.
Time Frame: Baseline through Month 12, Month 18, Month 24, and Month 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
percentage of participants
  Month 12 | 90 [55.5 to 99.7]
  Month 18 | 80 [44.4 to 97.5]
  Month 24 | 80 [44.4 to 97.5]
  Month 36: number analyzed (Participants) | 8
  Month 36 | 75 [34.9 to 96.8]

3. Secondary Outcome: Median Age At Death
Description: Age at death for participants who died during the study. All deaths were assessed by the Investigator as unrelated to study drug.
Time Frame: Baseline through Month 36
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 2
months | 9.33 [4.9 to 13.8]

4. Secondary Outcome: Change From Baseline In Percentiles For Weight For Age (WFA) At 12, 24, And 36 Months
Description: This outcome measure evaluated the effects of sebelipase alfa on growth by measuring the changes from baseline in percentiles for WFA. Percentiles for WFA were summarized as observed values by visit. Baseline was defined as the last available assessment prior to the first infusion of sebelipase alfa.
Time Frame: Baseline, Month 12, Month 24, and Month 36
Population: as for outcome 1
Measure: Median (Full Range); unit: percentile
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 9
percentile
  Month 12: number analyzed (Participants) | 8
  Month 12 | 27.760 [1.34 to 67.58]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 41.276 [7.54 to 63.77]
  Month 36: number analyzed (Participants) | 5
  Month 36 | 59.310 [36.39 to 72.51]

5. Secondary Outcome: Number Of Participants With Stunting, Wasting, Or Underweight At Baseline, 12, 24, And 36 Months
Description: The number of participants who met criteria for the following 3 dichotomous indicators of under nutrition were reported. These indicators included the following:
  1. Stunting was defined as at least 2 standard deviations below the median for length-for-age/height-for-age.
  2. Wasting was defined as wasting at least 2 standard deviations below the median for weight-for-length/weight-for-height.
  3. Underweight was defined as at least 2 standard deviations below the median for WFA.
Time Frame: Baseline to Month 12, Month 24, and Month 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
Participants
  Stunting, Baseline: number analyzed (Participants) | 9
  Stunting, Baseline | 4
  Stunting, Month 12: number analyzed (Participants) | 8
  Stunting, Month 12 | 0
  Stunting, Month 24: number analyzed (Participants) | 8
  Stunting, Month 24 | 0
  Stunting, Month 36: number analyzed (Participants) | 5
  Stunting, Month 36 | 0
  Wasting, Baseline: number analyzed (Participants) | 9
  Wasting, Baseline | 5
  Wasting, Month 12: number analyzed (Participants) | 8
  Wasting, Month 12 | 0
  Wasting, Month 24: number analyzed (Participants) | 8
  Wasting, Month 24 | 0
  Wasting, Month 36: number analyzed (Participants) | 5
  Wasting, Month 36 | 0
  Underweight, Baseline | 6
  Underweight, Month 12: number analyzed (Participants) | 8
  Underweight, Month 12 | 0
  Underweight, Month 24: number analyzed (Participants) | 8
  Underweight, Month 24 | 0
  Underweight, Month 36: number analyzed (Participants) | 5
  Underweight, Month 36 | 0

6. Secondary Outcome: Change From Baseline In Serum Transaminases (ALT And AST) At Month 12, 24, And 36
Description: This outcome measure evaluated the effects of sebelipase alfa on liver function by measuring the change from baseline in alanine aminotransferase (ALT) and aspartate aminotransferase (AST) at months 12, 24, and 36. Results are reported in units/liter (U/L).
Time Frame: Baseline, Month 12, Month 24, and Month 36
Population: as for outcome 1
Measure: Median (Full Range); unit: U/L
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
U/L
  ALT: Month 12: number analyzed (Participants) | 7
  ALT: Month 12 | 0 [-175 to 66]
  ALT: Month 24: number analyzed (Participants) | 7
  ALT: Month 24 | 14.0 [-207 to 80]
  ALT: Month 36: number analyzed (Participants) | 4
  ALT: Month 36 | -42.0 [-224 to 6]
  AST: Month 12: number analyzed (Participants) | 6
  AST: Month 12 | -33.5 [-322 to 8]
  AST: Month 24: number analyzed (Participants) | 5
  AST: Month 24 | -4.0 [-90 to 36]
  AST: Month 36: number analyzed (Participants) | 3
  AST: Month 36 | -101.0 [-351 to -9]

7. Secondary Outcome: Change From Baseline In Serum Ferritin At Month 12, 24, And 36
Description: The median change in the inflammatory marker serum ferritin from Baseline to Months 12, 24, and 36 is presented. The number of participants analyzed reflects only those from the FAS who had both a baseline value and a value at the indicated timepoint (Months 12, 24, and 36). Results are reported in micrograms (ug)/L.
Time Frame: Baseline, Month 12, Month 24, and Month 36
Population: as for outcome 1
Measure: Median (Full Range); unit: ug/L
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 2
ug/L
  Month 12: number analyzed (Participants) | 1
  Month 12 | -2957.00 [-2957.0 to -2957.0]
  Month 24 | -1722.00 [-2984.0 to -460.0]
  Month 36: number analyzed (Participants) | 0

8. Secondary Outcome: Number Of Participants Achieving And Maintaining Transfusion-free Hemoglobin Normalization (TFHN)
Description: The number of participants achieving and maintaining TFHN are presented. For TFHN to be achieved, the participant had to meet the following criteria:
  1. Two post baseline measurements of hemoglobin, at least 4 weeks apart, were above the age-adjusted lower limit of normal (LLN);
  2. No known additional measurements of hemoglobin were below the age-adjusted LLN during the (minimum) 4 week period;
  3. No transfusions were administered to the participant during the (minimum) 4 week period, or for 2 weeks prior to the first hemoglobin measurement in the (minimum) 4 week period. If all 3 criteria were met, a participant was considered to have achieved TFHN on the date of the first hemoglobin assessment in the 4 week period. A participant was considered to have maintained TFHN if he/she was transfusion free at Week 6 and had no abnormally low hemoglobin levels (levels below the age adjusted LLN) beginning at Week 8 of the study and continuing for at least 13 weeks (3 months).
Time Frame: Baseline through Month 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 10
Participants
  Achieved TFHN | 7
  Maintained TFHN | 0

ADVERSE EVENTS:
Time Frame: Screening (up to 21 days prior to start of treatment) to Month 37 (approximately 30 days after the last dose of study drug).
Groups:
- Sebelipase Alfa: 1.0 mg/kg qw: This reporting group is based on the FAS and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 1.0 mg/kg qw. All 10 participants in the FAS received sebelipase alfa at a dose of 1.0 mg/kg qw.
- Sebelipase Alfa: 3.0 mg/kg qw: This reporting group is based on the FAS and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 3.0 mg/kg qw. Nine of the 10 participants in the FAS received sebelipase alfa at a dose of 3.0 mg/kg qw.
- Sebelipase Alfa: 5.0 mg/kg qw: This reporting group is based on the FAS and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 5.0 mg/kg qw. Seven of the 10 participants in the FAS received sebelipase alfa at a dose of 5.0 mg/kg qw.
- Sebelipase Alfa: 7.5 mg/kg qw: This reporting group is based on the FAS and includes AEs with onset during the administration of IV treatment of sebelipase alfa at a dose of 7.5 mg/kg qw (UK only). One of the 10 participants in the FAS received sebelipase alfa at a dose of 7.5 mg/kg qw.
Arm/Group | Sebelipase Alfa: 1.0 mg/kg qw | Sebelipase Alfa: 3.0 mg/kg qw | Sebelipase Alfa: 5.0 mg/kg qw | Sebelipase Alfa: 7.5 mg/kg qw
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/9 | 1/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 8/10 | 8/9 | 7/7 | 1/1
Other Adverse Events (participants affected / at risk) | 9/10 | 9/9 | 7/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sebelipase Alfa: 1.0 mg/kg qw (N=10) | Sebelipase Alfa: 3.0 mg/kg qw (N=9) | Sebelipase Alfa: 5.0 mg/kg qw (N=7) | Sebelipase Alfa: 7.5 mg/kg qw (N=1)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (5) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The single occurrence of pericardial effusion in the 1.0 mg/kg qw group lead to death and was assessed by the Investigator as unrelated to study drug.
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 5 (8) | 4 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 6 (12) | 3 (4) | 1 (2)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 6 (7) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) — The single occurrence of sepsis in the 5.0 mg/kg qw group lead to death and was assessed by the Investigator as unrelated to study drug.
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abscess bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0/5 (0) | 0/5 (0) | 1/4 (1) | 0/0 (0) — Only male participants were exposed to this adverse event
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug specific antibody present (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Body temperature fluctuation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sapovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embedded device (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor venous access (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Bloody discharge (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sebelipase Alfa: 1.0 mg/kg qw (N=10) | Sebelipase Alfa: 3.0 mg/kg qw (N=9) | Sebelipase Alfa: 5.0 mg/kg qw (N=7) | Sebelipase Alfa: 7.5 mg/kg qw (N=1)
Vomiting (Gastrointestinal disorders) | 5 (11) | 6 (15) | 4 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (12) | 5 (23) | 5 (29) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (5) | 2 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infantile spitting up (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (15) | 7 (43) | 5 (36) | 1 (5)
Pain (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (3) | 1 (1) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Catheter site discharge (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site extravasation (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Catheter site granuloma (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrophy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypochromasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node calcification (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 4 (5) | 2 (5) | 1 (1)
Device related sepsis (Infections and infestations) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 4 (8) | 2 (7) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 4 (4) | 1 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (4) | 2 (2) | 2 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 3 (3) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Parainfluenza virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ctyomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis sapovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Parechovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (2) | 1 (4) | 0 (0)
Heart rate increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Vitamin E decreased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 1 (2) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Body temperature abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Drug specific antibody present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Alpha 1 foetoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alpha-1 anti-trypsin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Antibody test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Beta-2 glycoprotein antibody (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood aldosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood aldosterone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood parathyroid hormone (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure abnormal (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brucella test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 1 (3) | 1 (5) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug specific antibody (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecal calprotectin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric fluid analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasogastric output abnormal (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Norovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osmolar gap increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parvovirus B19 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin level decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin A decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyposideraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin A deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin E deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 3 (4) | 4 (4) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device infusion issue (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 4 (19) | 4 (8) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (6) | 4 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (8) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (9) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 2 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 1 (3) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 5 (8) | 6 (13) | 3 (5) | 1 (3)
Bradycardia (Cardiac disorders) | 3 (4) | 2 (2) | 2 (3) | 0 (0)
Cardiac septal hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphodema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microangiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site extravasation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eyelid rash (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staring (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chimerism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromosomal deletion (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic calcification (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/5 (0) | 0/4 (0) | 1/3 (1) | 0 (0) — Only female participants were exposed to this adverse event
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (4) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02193867/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT02193867/SAP_001.pdf